CLINICAL TRIAL: NCT03180203
Title: The Full Closed Loop Ventilation Mode INTELLiVENT-ASV: User-friendly and Effective Mechanical Ventilation in High Risk Postoperative Patient on the Intensive Care Unit
Brief Title: Postoperative INTELLiVENT-ASV Ventilation
Acronym: POSITiVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Ashley De Bie, MSc., Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL58975.100.16
Record Dates: First submitted 2017-05-30; First posted 2017-06-08 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Ventilators, Mechanical; Intensive Care Units; Postoperative Care
Keywords: INTELLiVENT-ASV; Fully closed-loop ventilation; Wean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The participant will not know which ventilation mode will be or is used. The primairy investigator and care providers are aware of which ventilation mode is used since it is not possible to blind the care providers because they will need to change ventilating parameters if necessary.
  The outcome assesor for the percentages of time will be masked. Also are the radiologists, who judge the postoperative thoracic x-ray, masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTELLiVENT-ASV (Experimental): INTELLiVENT-ASV is a full closed-loop ventilation mode,available on the mechanical ventilator S1 of Hamilton.
  Interventions: Device: INTELLiVENT-ASV
- Conventional modes (Active Comparator): Volume controlled continuous mandatory ventilation (CMV) mode with pressure support mode on the Hamilton S1 Device.
  Interventions: Device: Conventional modes

INTERVENTIONS:
Device: INTELLiVENT-ASV — After ICU admission:
  * The first three hours: only ventilation with INTELLiVENT-ASV with Quickwean.
  * After three hours: Automatic spontaneous breathing trials (SBT) is activated and SBT starts if >10minutes PEEP:<9cmH2O,FiO2:<41%,VT/IBW<5ml/kg and RSB:<106l/l*min.
  Settings SBT are MV% 25%,PEEP 5cmH2O.SBT automatically stops if respiratory rate >35b/min or increases >100% since start of SBT, FiO2 >50%, PeTCO2 increases >8mmHg.
  Extubation criteria: Leakage <50ml/hr,hemodynamically stable, awake with enough muscle strength and successful SBT >10min.
  If during mechanical ventilation the ICU care providers decide that it is necessary for the treatment, they may switch to another ventilation mode or extubate without a SBT.
  Arms: INTELLiVENT-ASV
Device: Conventional modes — After ICU admission:
  The first three hours: only ventilation with CMV or PS. If required care providers may change the mode to adaptive support ventilation.
  After three hours: manual SBT is required if >10min PS<11cmH2O,PEEP<9cmH2O,FiO2<41%.
  Settings SBT are PS 5cmH2O, PEEP 5cmH2O, FiO2 30%. SBT must be stopped if respiratory rate >35b/min or increases >100% since the start of SBT, saturation <92% or the PeTCO2 increases >8mmHg.
  Extubation criteria: Leakage <50ml/hr,hemodynamically stable, awake with enough muscle strength and successful SBT >10min.
  If during mechanical ventilation the ICU care providers decide that it is necessary for the treatment, they may switch to another ventilation mode or extubate without a SBT.
  Arms: Conventional modes

SUMMARY:
The aim of this study is to investigate whether postoperative ventilation with INTELLiVENT-ASV(adaptive support ventilation) in high risk patients, after cardiothoracic surgery, is as effective, more user-friendly and as safe as compared to the conventional modes of ventilation.

DETAILED DESCRIPTION:
Recently, Hamilton Medical has introduced the new mechanical ventilation mode "INTELLiVENT-ASV". This is a fully closed ventilation mode that can automatically adjust the ventilation settings based on the measured End tidal CO2 (ETCO2) and the measured saturation (SpO2) in both passive and active ventilated patients. Current literature has shown that this mode is safe to use in patients admitted on the intensive care unit. A pilot study in the Catharina Hospital Eindhoven confirmed that in postoperative low risk patients on the intensive care unit INTELLiVENT-ASV is safe. Compared to continuous mandatory or pressure controlled ventilation with pressure support (conventional mechanical ventilation), INTELLiVENT-ASV is even as effective as conventional mechanical ventilation, with a significantly reduced number of interactions with the ventilator. However, available research about the effectiveness of INTELLiVENT-ASV in postoperative high risk patients is lacking. Also the knowledge about the user-friendliness of the above modes of mechanical ventilation for the users is lacking.

This is a prospective randomized study with a control group and a intervention group of postoperative high risk patients. Through randomization will be determined whether the participant, after surgery, will be mechanically ventilated with INTELLiVENT-ASV and Quickwean or with conventional mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years of age.
* Informed consent.
* Body mass index of <35 kg/m2.
* Mechanical ventilation after elective cardiothoracic surgery.
* Admission of the patient after surgery is on the high care unit of the intensive care ward for postoperative mechanical ventilation.

Exclusion Criteria:

* Withdrawal of consent
* Medical history of a pneumonectomy or lobectomy.
* The patient wit acute respiratory distress syndrome after surgery.
* The patient with a medical history of COPD Gold 3 or 4.
* The patient is participating in another postoperative study performed on the intensive care.
* The patient is, preoperatively determined, eligible for a fast-track postoperative treatment program on the Post Anesthesia Care Unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of mechanical ventilation time in an optimal, acceptable or unacceptable ventilation zone. | During the first 3 hours, since admission on the ICU with the start of the intervention ventilation mode.
  * An optimal zone = Tidal volume (TV) = 4-8 ml/kg of the predicted body weight (PBW) with an EtCO2 = 30-45mmHg, a plateau pressure = <31cmH2O and SpO2 = 93-98%.
  * An acceptable zone = TV = 8-12 ml/kg of PBW with an EtCO2 = 25-30 or 45-50mmHg, a plateau pressure = 31-35 cmH2O and SpO2 = 85-93% or >98%.
  * An unacceptable zone = TV >12 ml/kg of PBW or an EtCO2 = <25 or >50mmHg, plateau pressure >35 cmH2O or SpO2 = <85%.

SECONDARY OUTCOMES:
The percentage (%) of successful extubations. | During the first 24, 48 and 72 hours after extubation
  A successful extubation is an extubation without a new intubation or the use of non-invasive ventilation within 24, 48 or 72 hours.
Postoperative weaning time | 72 hours
  The time from admission on the ICU and a temperature of >35.5°C until extubation.
Workload | 72 hours
  The number of alarms and required interactions between the ventilator and the user during mechanical ventilation on the ICU.
Usability | Up to 1 day after extubation
  A survey with acceptance score (1-10) completed by the care provider at the bedside who treated the patient for the weaning
Patient agitation | Up to 72 hours of mechanical ventilation time
  The number of agitated moments of the patient recognized by the ICU care provider at the bedside.
Administration of sedatives and analgesics | Up to 72 hours of mechanical ventilation time
  The number and dosages of administrations of NSAIDs, opiates, benzodiazepines, clonidine, propofol or haloperidol during mechanical ventilation.
The Richmond Agitation-Sedation Scale (RASS) | Up to 72 hours of mechanical ventilation time
  The RASS for every hour during mechanical ventilation.
Postoperative atelectasis | Up to 48 hours after extubation
  The number of a patients with an atelectasis on the first thoracic x-ray or the thoracic x-ray the following day after surgery.
CO2 levels for postoperative pulmonary shunting | Up to 72 hours of mechanical ventilation time
  The EtCO2/pCO2 ratio during mechanical ventilation.
O2 levels for postoperative pulmonary shunting | Up to 72 hours of mechanical ventilation time
  The pO2/FiO2 ratio during mechanical ventilation.
Reliability of non-invasive oxygen saturation measurement | 72 hours
  The time of mechanical ventilation on the ICU without non-invasive measurement of the oxygen saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley De Bie Dekker, Msc, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beijers AJ, Roos AN, Bindels AJ. Fully automated closed-loop ventilation is safe and effective in post-cardiac surgery patients. Intensive Care Med. 2014 May;40(5):752-3. doi: 10.1007/s00134-014-3234-7. Epub 2014 Feb 28. No abstract available. PMID 24577110
- [Background] Lellouche F, Bouchard PA, Simard S, L'Her E, Wysocki M. Evaluation of fully automated ventilation: a randomized controlled study in post-cardiac surgery patients. Intensive Care Med. 2013 Mar;39(3):463-71. doi: 10.1007/s00134-012-2799-2. Epub 2013 Jan 22. PMID 23338569
- [Derived] De Bie AJR, Neto AS, van Meenen DM, Bouwman AR, Roos AN, Lameijer JR, Korsten EHM, Schultz MJ, Bindels AJGH. Fully automated postoperative ventilation in cardiac surgery patients: a randomised clinical trial. Br J Anaesth. 2020 Nov;125(5):739-749. doi: 10.1016/j.bja.2020.06.037. Epub 2020 Jul 30. PMID 32739044
- Available data/document: Study Protocol: Study Intensive Care — https://www.catharinaziekenhuis.nl/contact.html — Contact can be made to request the study protocol (Dutch)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT03180203/Prot_SAP_001.pdf